CLINICAL TRIAL: NCT02205515
Title: An Open Label, Single-Centre, Pilot Study for Radiosensitization of Everolimus With External Beam Radiotherapy for the Treatment of Metastatic Neuroendocrine Liver Metastasis
Brief Title: An Open Label, Single-Centre, Pilot Study of Everolimus With EBRT for the Treatment of mNET Liver Metastasis
Acronym: EBRT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: File#13-907/OZM-057
Record Dates: First submitted 2014-06-25; First posted 2014-07-31 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Carcinoma, Neuroendocrine
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Other): SBRT or EBRT
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Everolimus is a novel derivative of rapamycin.
  Other Names: Afinitor

SUMMARY:
Approximately 50% of patients with neuroendocrine cancers present with metastasis, a vast majority to the liver. In such patients, one treatment option for liver-directed therapy is surgical resection. However, a significant proportion of patients are not eligible for resection because of patient factors (age, comorbidities) or tumor-related factors.

There have been scant data on the utility of EBRT (external-beam radiotherapy) and SABR (stereotactic ablative radiotherapy) for metastatic neuroendocrine tumors of the liver. This study will measure the effects of concurrent everolimus with external-beam radiotherapy to the liver for metastatic neuroendocrine New methods of tumor assessment are needed in NETs. Three new techniques are being developed at the Sunnybrook Research Institute to assess tumour response to treatment: (1) contrast enhanced ultrasound; (2) perfusion CT; and (3) perfusion MRI. These methods are devised to measure tumour perfusion and blood flow as response indicators and can measure cell death non-invasively.

1. Concurrent everolimus given with external-beam radiotherapy to the liver for metastatic neuroendocrine tumors of the liver will enhance the efficacy of radiotherapy and add little, if any, toxicity
2. New radiological measures of CEUS and DCE-CT are effective measure to delineate tumor response in NETs.

DETAILED DESCRIPTION:
This is an open label, single-centre, pilot study for Radiosensitization of Everolimus with external beam radiotherapy to the liver for metastatic neuroendocrine tumors The study will have 2 safety run-in dose levels: 2.5mg and 5mg Everolimus PO daily. Two patients will be enrolled into the 2.5mg dose level and 2 patients enrolled into the 5mg dose level. However, only one patient can start the safety run-in doses at a time. For the safety run-in dose levels, if no serious adverse events related to Everolimus occur within 30 days of the first dose of radiation therapy (in combination with Everolimus) in one patient, then the next patient can start study drug. The same criteria applies for the first 4 patients (2 patients on 2.5mg PO daily and 2 patients on 5 mg PO daily).

If no serious adverse events related to Everolimus occur in the fourth patient at 5mg PO daily within 30 days of the first dose of radiation therapy (in combination with Everolimus), more than one patient can then be enrolled at one time at the target dose of 7.5mg PO daily. Ten patients will be enrolled at 7.5mg PO daily.

For all patients, Everolimus starts 30 days prior to radiation and continues throughout radiation and for 14 days post radiation. Patients will receive Everolimus for 14 days post treatment only; as this pilot is designed to assess the combined effect of radiation and Everolimus.

All patients will receive external-beam radiotherapy (30Gy in 10 fractions) or SBRT (up to 60Gy in 3-5 fractions given on alternating weekdays over 1-2 weeks). The decision to treat with either external-beam radiotherapy or SBRT will be based on whether the lesions are amenable to SBRT (preferred treatment), which is determined by the size of the target lesion, liver sparing and organs-at-risk dose constraints. The prescription dose of external-beam radiotherapy and SBRT will similarly be determined by these factors.

ELIGIBILITY:
Inclusion Criteria:

1. Histological and/or cytological diagnosis of unresectable neuroendocrine tumor with liver metastases confirmed on imaging scans
2. Ki-67<55%
3. No prior Everolimus within 3 months prior to registration
4. No prior radiotherapy to the liver
5. 1-3 liver metastatic lesions confirmed on imaging scans
6. Size of target metastatic lesion is 6 cm or less
7. At least 700 cc of liver uninvolved by tumor
8. Previous liver resection, systemic therapy or local ablation therapy (radiofrequency ablation, transarterial chemoemolization, radioemolization) is allowed.
9. Extrahepatic disease is allowed if maximum involved organs (including the liver) is 3 or less (i.e. oligometastases).
10. Child-Pugh's A liver function
11. Male or female: Age ≥ 18 years
12. Life expectancy > 6 months
13. ECOG PS ≤1
14. Laboratory Requirements - within 14 days prior to registration:

    Hematology Absolute Neutrophils Count ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L Hemoglobin ≥ 90 g/L Biochemistry Serum Bilirubin ≤ 1.5 x upper limit of normal Serum Creatinine ≤ 1.5 x upper limit of normal AST ≤ 3 x upper limit of normal ALT ≤ 3 x upper limit of normal INR ≤ 1.5 Fasting Serum Cholesterol ≤ 300 mg/dl or 7.75 mmol/L Fasting Triglycerides ≤ 2.5 x ULN Adequate Glucose Control Urinalysis Proteinuria ≤ grade 1 (by dipstick)
15. Before patient registration/randomization, written informed consent must be given according to local Institutional and/or University Human Experimentation Committee requirements. The patient must sign the consent form prior to randomization or registration.
16. Patients that have a positive HBV-DNA result at screening must agree to take prophylactic treatment for 1-2 weeks prior to beginning Everolimus treatment. See section 7.2 for further information on Viral Hepatitis management
17. Patients must be accessible for treatment and follow-up. Patients registered on this trial must be treated and followed at the participating centre. Investigators must assure themselves the patients registered on this trial will be available for complete documentation of the treatment, adverse events response assessment and follow-up.

Exclusion Criteria:

1. Major surgical procedure, open biopsy or significant traumatic injury within 28 days prior to registration (i.e. patients must have recovered to less than or equal to grade 1 from any major surgery), or anticipation of need for major surgical procedure during or within 7 weeks after chemo-radiotherapy
2. Known to have clinical or radiological evidence of CNS metastases
3. Patients with hepatitis
4. Patients with neuroendocrine tumor of a pancreatic origin
5. Patients with a past or current history (within last 2 years) of other malignancies, except for the indication under this study and curatively treated basal and squamous skin cancer or in-situ cancer of the cervix. Prior treatment of localized prostate cancer is permitted if treatment was greater than 5 years ago and the patient currently has no biochemical evidence of recurrence.
6. Uncontrolled diabetes mellitus
7. Active bleeding diathesis, or an oral anti-vitamin K medication (except low dose warfarin, LMWH, or acetylsalicylic acid or equivalent) as long as the INR is <1.5.
8. Patients with known history or present encephalopathy
9. Gross clinically detectable ascites
10. Any comorbidity or concomitant medication that would contraindicate treatment with Everolimus
11. Women of childbearing potential with a positive pregnancy test at baseline or lactating. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Females patients must not be pregnant or become pregnant during this study and for 6 months after the last dose of Everolimus
12. Sexually active males and females (of childbearing potential) unwilling to practice contraception during the study. Patients of childbearing potential must be willing to use a reliable method of birth control. i.e.: double barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device or tubal ligation during the study.
13. Prior radiotherapy to the right upper quadrant of the liver
14. Contraindication to CT dye injection
15. Contraindication to MRI
16. Contraindication to CEUS dye injection
17. Body habitus and or tumor location not allowing for CEUS
18. Any other serious intercurrent illness such as cardiovascular disease, HIV or any neurological disease
19. Patients taking other approved or investigational drug/anticancer treatment (other than ongoing androgen ablation and oral prednisone which are permitted) during the study period, including chemotherapy, biological response modifiers, immunotherapy, surgery or radiotherapy.
20. Patients concurrently participating in another clinical trial
21. Patients unwilling to or unable to comply with the treatment plan
22. Patients who have metastatic liver lesions that are candidates for resection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03; Primary Completion 2021-09 (Actual); Study Completion 2021-10 (Actual)

PRIMARY OUTCOMES:
The tolerability and efficacy of Everolimus concurrent with external-beam radiotherapy will be examined | Through study completion an average of 1 year

SECONDARY OUTCOMES:
The response rate (as measured by RECIST version 1.1 criteria) of combined treatment with Everolimus and radiation to metastatic liver lesions in neuroendocrine cancers will be examined | Screening, every 12weeks during the study until off-treatment due to progression
The association between tumor perfusion and blood flow in vivo as measured by dynamic contrast-enhanced (DCE)-CT, CEUS, with clinical safety and efficacy outcomes will be preliminary explored | During the duration of the study
The effects of tumor perfusion and blood flow (on liver metastasis) as measured by DCE-MRI, DCE-CT and CEUS at baseline, during Everolimus but prior to SBRT, and post-SBRT in patients with neuroendocrine cancer metastatic to liver will be explored | Screening, Day 26-28, and 7 days follow-up after last RT
The biochemical response (Urinary 5HIAA and Chromogranin A) of combined treatment with Everolimus and radiation to metastatic liver lesions in neuroendocrine cancers will be examined | Screening, Day 26-28, and 7 days follow-up after last RT, 30 & 90 days after completing radiotherapy and at progression. 5HIAA to be also done as clinically indicated

CONTACTS AND LOCATIONS:
Overall Officials: Simron Singh, MD, Principal Investigator — Odette Cancer Centre, Sunnybrook HSC
Locations (1):
- Odette Cancer Centre, Sunnybrook Health Science Centre, Toronto, Ontario, Canada